CLINICAL TRIAL: NCT04806906
Title: A Phase 2, Monocentric, Pilot Study to Evaluate Safety and Efficacy of CC 486 (Oral Azacitidine) Plus Best Supportive Care as Maintenance of Response to sc Azacitidine in IPSS Higher Risk Elderly MDS Patients
Brief Title: Pilot Study of CC 486 (Oral Azacitidine) Plus BSC as Maintenance After sc Azacitidine in Elderly HR-IPSS-R MDS Patients
Acronym: FLO_CC-486-
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florence (Other)
Responsible Party: Principal Investigator, Valeria Santini, Professor, University of Florence
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: University of Florence
Record Dates: First submitted 2021-02-23; First posted 2021-03-19 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: MDS; CMML
Keywords: Azacitidine; Therapy; DNA methylation analysis
MeSH Terms: interventions — cc-486; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CC-486 (Experimental): subjects will receive 300 mg CC-486 QD for 14 days of each 28-day treatment cycle
  Interventions: Drug: CC-486

INTERVENTIONS:
Drug: CC-486 — Investigational product will be dispensed on Day 1 of each treatment cycle. 300 mg CC-486 QD for 14 days of each 28-day treatment cycle
  Other Names: Oral Azacitidine

SUMMARY:
Treatment of higher-risk (intermediate, high and very high) Myelodysplastic Syndromes (MDS) according to the revised International Prognostic Scoring System (IPSS-R) who obtained a stable hematological response ( CR, PR) after subcutaneous azacitidine treatment.

Azacitidine is administered in hospital in a day care regimen, in Italy only by subcutaneous injection. The long duration of therapy obliges patients to travel to the hospital regularly, with evident worsening quality of life, both for patients and caregivers, although balanced by prolongation of survival and hematological improvement. Many patients stop therapy or are reluctant to continue because of the dependence from caregivers and hospital care.

This clinical study will evaluate the efficacy and safety of oral azacitidine (CC-486) plus best supportive care in subjects with higher-risk (intermediate, high and very high) Myelodysplastic Syndrome (MDS) according to the revised International Prognostic Scoring System (IPSS-R) and (high and INT-2) according to IPSS who obtained a stable hematological response (CR, PR, SD with HI) after at least 4-6 cycles of subcutaneous azacitidine treatment and maintained for 2 additional cycles.

DETAILED DESCRIPTION:
Azacitidine therapy is effective in prolonging survival in higher risk MDS patients provided therapy is administered at 28 day-cycles until progression or loss of response.

A study conducted several years ago shows that although most responses to azacitidine occurred within 6 cycles, continued azacitidine therapy led to a further improvement in response category in almost half (48%) of all responders with a median of 3 additional cycles, and that 92% of patients achieved their best response by Cycle 12. In a randomized phase 3 trial conducted by the US Cancer and Leukemia Group B, which compared azacitidine with best supportive care, most responses occurred during the third or fourth month of azacitidine therapy. The phase 3 Cancer and Leukemia Group B study also showed that 90% of responses occurred within the first 6 cycles of treatment and that best response generally occurred 2 cycles after the first response-all of which is consistent with the current findings. Taken together, these data suggest that although some effects of azacitidine manifest promptly, additional courses are usually necessary before best response is achieved. Therefore, continuing azacitidine therapy offers the best chance of enhanced benefit if treatment is tolerated and there is no evidence of disease progression.

Azacitidine may affect the differentiation and growth of the MDS clone without necessarily eradicating it, suggesting that repetitive and prolonged exposure to azacitidine may be necessary for both the initial effects and the subsequent augmentation of response. Discontinuation of azacitidine therapy is in fact invariably followed by loss of response, disease progression and short survival. Treatment should be optimized to deliver at least 6 cycles, and in responsive patients until progression. In clinical practice, however, AZA is often discontinued after few cycles. Prematurely interrupted therapy could be the cause of inferior outcomes registered in "real life" studies. This inconsistency may be due to differences in adherence to dose, schedule, and minimum number of cycles, as well as to the management of patients with severe comorbidities. Proper management of first-line azacitidine therapy, with appropriate doses and prolonged treatment, may partially reduce primary resistance. This is why it is extremely important to maintain treatment until progression, despite scarce compliance of the patients to subcutaneous injections. Anyhow, it is clear that the azacitidine effect is transient, with responses maintained for 6 to 24 months.

Survival of the patients with refractory/relapsed disease is extremely short. A premature arrest of treatment may thus provoke loss of response and accelerate progression. In order to improve the compliance to treatment of MDS patients who have shown optimal responses to azacitidine, an oral formulation of the drug could indeed be advantageous. Oral therapy with CC 486 could free patients from hospital and caregiver dependence, as well as from injection site reactions, consequently improving quality of life, without altering the necessary continuation of treatment. During the present Covid-19 outbreak it has became even clearer that treatment with medications in oral formulation, under strict control of treating physicians, may indeed, beyond improving quality of life, decrease the risk of exposure to infections derived by in hospital administered therapy for MDS patients.

An oral formulation of azacitidine like cc486 provides an opportunity to deliver the drug at lower systemic doses over a more prolonged schedule that can be practically achieved with parenteral therapy. In addition, an oral formulation that can be taken at home rather than in the hospital/clinic setting represents an opportunity for patients with MDS to have a more convenient route of administration, thus alleviating the morbidity of injection and avoiding the inconvenience and resource utilization costs associated with frequent hospital/clinic visits. In addition, intervention with azacitidine in patients with MDS that have obtained a response after sc azacitidine may offer better quality of life and possibly a survival advantage.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

1. Male or female subjects ≥ 65 years of age at the time of signing the ICD;
2. Diagnosed, histologically confirmed at inclusion,

   * Int-2 or High according to IPSS, or
   * Very High, High or Intermediate according to IPSS-R, or
   * Hypoplastic AML (20-30% BM blasts, previosuly considered MDS RAEB-T)
   * myelodysplastic CMML (included in IPSS scoring, WBC < 13.x 109/L);
3. Should have undergone therapy with subcutaneous azacitidine for at least 4-6 cycles ( + 2 cycles)
4. Must have achieved CR/CRi, PR or SD with HI status, as evidenced by IWG Criteria 2006 ( APPENDIX E):
5. ECOG performance status of 0, 1, 2 (Appendix C);
6. Adequate bone marrow function based on ANCs ≥ 1.0 x 109/L and platelet counts ≥ 70 x 109/L.
7. Adequate organ function, defined as:

Serum bilirubin ≤1.5 times the upper limit of normal (ULN); Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 times the ULN; Serum creatinine ≤ 2.5 times the ULN; 8.Male subjects with a female partner of childbearing potential must agree to practice abstinence or to the use of a physician-approved contraceptive method throughout the course of the study and avoid fathering a child during the course of the study and for 3 months following the last dose of azacitidine; 10. Understand and voluntarily sign an ICD prior to any study related assessments/procedures are conducted; 11. Able to adhere to the study visit schedule and other protocol requirements; 12. Ability to swallow study medication.

Exclusion Criteria:

* Absence of confirmed hematological response ( IWG HI/PR/CR) after at least 4 to 6 months of azacitidine sc and maintenance of response for 2 additional cycles.
* Inability to provide a valid informed consent.
* Eligibility for HSCT
* Active infection
* Serum creatinine > 2 x ULN at screening.
* ECOG performance status > 2
* Left ventricular ejection fraction < 50% by echocardiography
* A history of repeated hospitalization for severe infections Systemic diseases that would prevent study treatment (e.g. uncontrolled hypertension, cardiovascular, renal, hepatic, metabolic, etc.)
* Clinical or laboratory evidence of chronic Hepatitis B or Hepatitis C (definition of
* chronic hepatitis follows EASL 2017 criteria).
* History of HIV positive test result (ELISA or Western blot).
* ALT or AST over 3 times superior to ULN at screening.
* Total bilirubin over 1.5 times superior to ULN at screening (patients with Gilbert syndrome are allowed to enter the study)
* Patients participating in another clinical trial other than an observational registry study.
* Patients with a history of another malignancy within the past 3 years, with the exception of basal skin carcinoma or cervical carcinoma in situ or completely resected colonic polyps carcinoma in situ.
* History of non-compliance to medical regimens, or patients who are considered potentially unreliable and/or not cooperative.
* Presence of a surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of study drug.
* History of drug or alcohol abuse within the 12 months prior to enrollment.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 11 (Estimated)
Dates: Start 2021-03-24 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Maintenance or improvement of response to therapy after switching from sc azacitidine to (oral) CC-486 | 0-24 months
  Bone marrow aspirate will be performed before and after treatment, to evaluate maintenance of response according to IWG criteria. Assessment of complete and partial response, stable disease or progression will be provided by evaluating hematopoietic cell morphology. Routine interval of marrow assessments will be 4 months for safety. Marrow samples during treatment will be collected on Day 1 (± 7 days) every 4 cycles and at the Treatment Discontinuation visit. After Cycle 36, bone marrow aspiration collection and evaluation will occur if clinically indicated at the discretion of the Investigator. Additional bone marrow samples should be collected as clinically indicated. A bone marrow biopsy must be collected if adequate aspirate is not obtainable. Whenever a bone marrow sample is collected, a peripheral blood smear is to be prepared. Bone marrow cytogenetic testing by complete karyotype analysis is to be completed whenever a bone marrow aspirate is performed.
Safety and tolerability of cc 486 | 0-24 months
  Safety assessments will consist of evaluating adverse events and concomitant medication/therapies used to treat them, secondary primary malignancy, hematology and serum chemistry parameters, body weight measurement, vital signs, physical examinations, clinical signs and symptoms, with great attention to GI symptoms, laboratory, pathological, radiological or surgical findings and pregnancy testing (for FCBP subjects). Urinalysis and ECG will be repeated whenever clinically indicated during treatment and according routine HR-MDS patient management. Second primary malignancies will be monitored as events of interest and should be included as part of the assessment of AEs throughout the duration of the study including post treatment follow-up period. Investigators are to report any second primary malignancy, regardless of causal relationship to CC-486, occurring at any time from signing of informed consent and until the last study visit.
Patient reported outcome on health related quality of life during CC-486 treatment | 0-24 months
  The patients treated with CC-486 will receive the questionnaire EQ-5D (EQ-5D-3L), a standardized instrument measuring health outcome. It provides a simple descriptive profile and a single index value for health status. Original EQ-5D questionnaire has five dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) and three distinct levels of functioning within each aspect (no problems, some problems and extreme problems). Each item is rescaled so that a better response corresponds to a higher numerical value and better QoL. Transformation of raw scores into a 0-100 scale will be carried out to generate the standardized scores for each domain. The EQ-5D questionnaire should be completed prior to interaction with study personnel and prior to CC-486 administration on Day 1 of every Cycle. Exploratory QoL Questions (Physical Impairment Numeric Rating Scale) will also be utilized in this clinical trial (scale 0-100).

SECONDARY OUTCOMES:
Time to relapse from CR/CRi, PR or SD with HI | 0-24 months
  The number of months elapsed from beginning of CC486 treatment to loss of marrow response will be evaluated . The first assessment of bone marrow status for maintenance or loss of response (CR/CRi, PR and SD with HI) will occur at Cycle 4. If response is maintained or improved, subjects can continue on to Cycle 5 and beyond. Subjects will be further assessed for response status every 4 cycles and at the Treatment Discontinuation visit. Assessment of marrow response will be performed at the discretion of the investigator in case of alterations in blood counts or unexpected cytopenias.
Time to discontinuation of treatment | 0-24 months
  The number of months elapsed from beginning of CC486 treatment and its end wil be evaluated.
  Subjects will be discontinued from treatment when they meet the following criteria:
  Loss of response and/or progression to AML as demonstrated by bone marrow aspiration and peripheral blood counts Completion of study treatment Unacceptable toxicity
Overall survival | 0-60 months
  The number of months elapsed from beginning of CC486 treatment to death

OTHER OUTCOMES:
Exploratory Objectives: measure modifications of the pattern of DNA methylation levels ( by ERRBS technique) during cc 486 treatment as compared with those evaluated at the moment of cessation of azacitidine sc administration. | 0-24 months
  ERRBS-identified DNA differentially methylated regions (DMRs) at baseline, and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Valeria Santini, MD, Study Chair — University of Florence- AOU Careggi
Locations (1):
- AOU Careggi- University of Florence, Florence, Italy

REFERENCES:
- [Background] Arber DA, Orazi A, Hasserjian R, Thiele J, Borowitz MJ, Le Beau MM, Bloomfield CD, Cazzola M, Vardiman JW. The 2016 revision to the World Health Organization classification of myeloid neoplasms and acute leukemia. Blood. 2016 May 19;127(20):2391-405. doi: 10.1182/blood-2016-03-643544. Epub 2016 Apr 11. PMID 27069254
- [Background] Agrawal K, Das V, Vyas P, Hajduch M. Nucleosidic DNA demethylating epigenetic drugs - A comprehensive review from discovery to clinic. Pharmacol Ther. 2018 Aug;188:45-79. doi: 10.1016/j.pharmthera.2018.02.006. Epub 2018 Feb 15. PMID 29454856
- [Background] Bejar R, Stevenson KE, Caughey B, Lindsley RC, Mar BG, Stojanov P, Getz G, Steensma DP, Ritz J, Soiffer R, Antin JH, Alyea E, Armand P, Ho V, Koreth J, Neuberg D, Cutler CS, Ebert BL. Somatic mutations predict poor outcome in patients with myelodysplastic syndrome after hematopoietic stem-cell transplantation. J Clin Oncol. 2014 Sep 1;32(25):2691-8. doi: 10.1200/JCO.2013.52.3381. Epub 2014 Aug 4. PMID 25092778
- [Background] Bernal T, Martinez-Camblor P, Sanchez-Garcia J, Sanz G. Effectiveness of azacitidine for the treatment of higher-risk myelodysplastic syndromes in daily practice: the authors' reply. Leukemia. 2016 Mar;30(3):740-1. doi: 10.1038/leu.2015.339. Epub 2016 Jan 12. No abstract available. PMID 26754826
- [Background] Benson AB 3rd, Ajani JA, Catalano RB, Engelking C, Kornblau SM, Martenson JA Jr, McCallum R, Mitchell EP, O'Dorisio TM, Vokes EE, Wadler S. Recommended guidelines for the treatment of cancer treatment-induced diarrhea. J Clin Oncol. 2004 Jul 15;22(14):2918-26. doi: 10.1200/JCO.2004.04.132. PMID 15254061
- [Background] Cabrero M, Jabbour E, Ravandi F, Bohannan Z, Pierce S, Kantarjian HM, Garcia-Manero G. Discontinuation of hypomethylating agent therapy in patients with myelodysplastic syndromes or acute myelogenous leukemia in complete remission or partial response: retrospective analysis of survival after long-term follow-up. Leuk Res. 2015 May;39(5):520-4. doi: 10.1016/j.leukres.2015.03.006. Epub 2015 Mar 20. PMID 25828745
- [Background] Cheson BD, Greenberg PL, Bennett JM, Lowenberg B, Wijermans PW, Nimer SD, Pinto A, Beran M, de Witte TM, Stone RM, Mittelman M, Sanz GF, Gore SD, Schiffer CA, Kantarjian H. Clinical application and proposal for modification of the International Working Group (IWG) response criteria in myelodysplasia. Blood. 2006 Jul 15;108(2):419-25. doi: 10.1182/blood-2005-10-4149. Epub 2006 Apr 11. PMID 16609072
- [Background] Cogle CR, Scott BL, Boyd T, Garcia-Manero G. Oral Azacitidine (CC-486) for the Treatment of Myelodysplastic Syndromes and Acute Myeloid Leukemia. Oncologist. 2015 Dec;20(12):1404-12. doi: 10.1634/theoncologist.2015-0165. Epub 2015 Oct 13. PMID 26463870
- [Background] de Lima M, Oran B, Champlin RE, Papadopoulos EB, Giralt SA, Scott BL, William BM, Hetzer J, Laille E, Hubbell B, Skikne BS, Craddock C. CC-486 Maintenance after Stem Cell Transplantation in Patients with Acute Myeloid Leukemia or Myelodysplastic Syndromes. Biol Blood Marrow Transplant. 2018 Oct;24(10):2017-2024. doi: 10.1016/j.bbmt.2018.06.016. Epub 2018 Jun 20. PMID 29933073
- [Background] Diesch J, Zwick A, Garz AK, Palau A, Buschbeck M, Gotze KS. A clinical-molecular update on azanucleoside-based therapy for the treatment of hematologic cancers. Clin Epigenetics. 2016 Jun 21;8:71. doi: 10.1186/s13148-016-0237-y. eCollection 2016. PMID 27330573
- [Background] Dinmohamed AG, van Norden Y, Visser O, Posthuma EF, Huijgens PC, Sonneveld P, van de Loosdrecht AA, Jongen-Lavrencic M. Effectiveness of azacitidine for the treatment of higher-risk myelodysplastic syndromes in daily practice: results from the Dutch population-based PHAROS MDS registry. Leukemia. 2015 Dec;29(12):2449-51. doi: 10.1038/leu.2015.220. Epub 2015 Sep 15. No abstract available. PMID 26369829
- [Background] Duong VH, Lin K, Reljic T, Kumar A, Al Ali NH, Lancet JE, List AF, Komrokji RS. Poor outcome of patients with myelodysplastic syndrome after azacitidine treatment failure. Clin Lymphoma Myeloma Leuk. 2013 Dec;13(6):711-5. doi: 10.1016/j.clml.2013.07.007. Epub 2013 Sep 17. PMID 24054159
- [Background] Fenaux P, Mufti GJ, Hellstrom-Lindberg E, Santini V, Finelli C, Giagounidis A, Schoch R, Gattermann N, Sanz G, List A, Gore SD, Seymour JF, Bennett JM, Byrd J, Backstrom J, Zimmerman L, McKenzie D, Beach C, Silverman LR; International Vidaza High-Risk MDS Survival Study Group. Efficacy of azacitidine compared with that of conventional care regimens in the treatment of higher-risk myelodysplastic syndromes: a randomised, open-label, phase III study. Lancet Oncol. 2009 Mar;10(3):223-32. doi: 10.1016/S1470-2045(09)70003-8. Epub 2009 Feb 21. PMID 19230772
- [Background] Fenaux P, Bowen D, Gattermann N, Hellstrom-Lindberg E, Hofmann WK, Pfeilstocker M, Sanz G, Santini V. Practical use of azacitidine in higher-risk myelodysplastic syndromes: an expert panel opinion. Leuk Res. 2010 Nov;34(11):1410-6. doi: 10.1016/j.leukres.2010.05.021. Epub 2010 Jul 6. PMID 20609474
- [Background] Figueroa ME, Skrabanek L, Li Y, Jiemjit A, Fandy TE, Paietta E, Fernandez H, Tallman MS, Greally JM, Carraway H, Licht JD, Gore SD, Melnick A. MDS and secondary AML display unique patterns and abundance of aberrant DNA methylation. Blood. 2009 Oct 15;114(16):3448-58. doi: 10.1182/blood-2009-01-200519. Epub 2009 Aug 3. PMID 19652201
- [Background] Gangat N, Patnaik MM, Begna K, Al-Kali A, Litzow MR, Ketterling RP, Hanson CA, Pardanani AD, Tefferi A. Survival trends in primary myelodysplastic syndromes: a comparative analysis of 1000 patients by year of diagnosis and treatment. Blood Cancer J. 2016 Apr 8;6(4):e414. doi: 10.1038/bcj.2016.23. No abstract available. PMID 27058229
- [Background] Garcia-Manero G, Stoltz ML, Ward MR, Kantarjian H, Sharma S. A pilot pharmacokinetic study of oral azacitidine. Leukemia. 2008 Sep;22(9):1680-4. doi: 10.1038/leu.2008.145. Epub 2008 Jun 12. PMID 18548103
- [Background] Garcia-Manero G, Gore SD, Cogle C, Ward R, Shi T, Macbeth KJ, Laille E, Giordano H, Sakoian S, Jabbour E, Kantarjian H, Skikne B. Phase I study of oral azacitidine in myelodysplastic syndromes, chronic myelomonocytic leukemia, and acute myeloid leukemia. J Clin Oncol. 2011 Jun 20;29(18):2521-7. doi: 10.1200/JCO.2010.34.4226. Epub 2011 May 16. PMID 21576646
- [Background] Garcia-Manero G, Gore SD, Kambhampati S, Scott B, Tefferi A, Cogle CR, Edenfield WJ, Hetzer J, Kumar K, Laille E, Shi T, MacBeth KJ, Skikne B. Efficacy and safety of extended dosing schedules of CC-486 (oral azacitidine) in patients with lower-risk myelodysplastic syndromes. Leukemia. 2016 Apr;30(4):889-96. doi: 10.1038/leu.2015.265. Epub 2015 Oct 7. PMID 26442612
- [Background] Garcia-Manero G, Almeida A, Giagounidis A, Platzbecker U, Garcia R, Voso MT, Larsen SR, Valcarcel D, Silverman LR, Skikne B, Santini V. Design and rationale of the QUAZAR Lower-Risk MDS (AZA-MDS-003) trial: a randomized phase 3 study of CC-486 (oral azacitidine) plus best supportive care vs placebo plus best supportive care in patients with IPSS lower-risk myelodysplastic syndromes and poor prognosis due to red blood cell transfusion-dependent anemia and thrombocytopenia. BMC Hematol. 2016 May 3;16:12. doi: 10.1186/s12878-016-0049-5. eCollection 2016. PMID 27148452
- [Background] Greenberg P, Cox C, LeBeau MM, Fenaux P, Morel P, Sanz G, Sanz M, Vallespi T, Hamblin T, Oscier D, Ohyashiki K, Toyama K, Aul C, Mufti G, Bennett J. International scoring system for evaluating prognosis in myelodysplastic syndromes. Blood. 1997 Mar 15;89(6):2079-88. PMID 9058730
- [Background] Greenberg PL, Tuechler H, Schanz J, Sanz G, Garcia-Manero G, Sole F, Bennett JM, Bowen D, Fenaux P, Dreyfus F, Kantarjian H, Kuendgen A, Levis A, Malcovati L, Cazzola M, Cermak J, Fonatsch C, Le Beau MM, Slovak ML, Krieger O, Luebbert M, Maciejewski J, Magalhaes SM, Miyazaki Y, Pfeilstocker M, Sekeres M, Sperr WR, Stauder R, Tauro S, Valent P, Vallespi T, van de Loosdrecht AA, Germing U, Haase D. Revised international prognostic scoring system for myelodysplastic syndromes. Blood. 2012 Sep 20;120(12):2454-65. doi: 10.1182/blood-2012-03-420489. Epub 2012 Jun 27. PMID 22740453
- [Background] Greenberg PL, Stone RM, Al-Kali A, Barta SK, Bejar R, Bennett JM, Carraway H, De Castro CM, Deeg HJ, DeZern AE, Fathi AT, Frankfurt O, Gaensler K, Garcia-Manero G, Griffiths EA, Head D, Horsfall R, Johnson RA, Juckett M, Klimek VM, Komrokji R, Kujawski LA, Maness LJ, O'Donnell MR, Pollyea DA, Shami PJ, Stein BL, Walker AR, Westervelt P, Zeidan A, Shead DA, Smith C. Myelodysplastic Syndromes, Version 2.2017, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2017 Jan;15(1):60-87. doi: 10.6004/jnccn.2017.0007. PMID 28040720
- [Background] Jabbour E, Garcia-Manero G, Batty N, Shan J, O'Brien S, Cortes J, Ravandi F, Issa JP, Kantarjian H. Outcome of patients with myelodysplastic syndrome after failure of decitabine therapy. Cancer. 2010 Aug 15;116(16):3830-4. doi: 10.1002/cncr.25247. PMID 20564137
- [Background] Jabbour EJ, Garcia-Manero G, Strati P, Mishra A, Al Ali NH, Padron E, Lancet J, Kadia T, Daver N, O'Brien S, Steensma DP, Sekeres MA, Gore SD, Dezern A, Roboz GJ, List AF, Kantarjian HM, Komrokji RS. Outcome of patients with low-risk and intermediate-1-risk myelodysplastic syndrome after hypomethylating agent failure: a report on behalf of the MDS Clinical Research Consortium. Cancer. 2015 Mar 15;121(6):876-82. doi: 10.1002/cncr.29145. Epub 2014 Nov 19. PMID 25410759
- [Background] Jiang Y, Dunbar A, Gondek LP, Mohan S, Rataul M, O'Keefe C, Sekeres M, Saunthararajah Y, Maciejewski JP. Aberrant DNA methylation is a dominant mechanism in MDS progression to AML. Blood. 2009 Feb 5;113(6):1315-25. doi: 10.1182/blood-2008-06-163246. Epub 2008 Oct 2. PMID 18832655
- [Background] Lee JH, Choi Y, Kim SD, Kim DY, Lee JH, Lee KH, Lee SM, Lee WS, Joo YD. Clinical outcome after failure of hypomethylating therapy for myelodysplastic syndrome. Eur J Haematol. 2015 Jun;94(6):546-53. doi: 10.1111/ejh.12469. Epub 2015 Jan 7. PMID 25315896
- [Background] Laille E, Shi T, Garcia-Manero G, Cogle CR, Gore SD, Hetzer J, Kumar K, Skikne B, MacBeth KJ. Pharmacokinetics and Pharmacodynamics with Extended Dosing of CC-486 in Patients with Hematologic Malignancies. PLoS One. 2015 Aug 21;10(8):e0135520. doi: 10.1371/journal.pone.0135520. eCollection 2015. PMID 26296092
- [Background] Malcovati L, Hellstrom-Lindberg E, Bowen D, Ades L, Cermak J, Del Canizo C, Della Porta MG, Fenaux P, Gattermann N, Germing U, Jansen JH, Mittelman M, Mufti G, Platzbecker U, Sanz GF, Selleslag D, Skov-Holm M, Stauder R, Symeonidis A, van de Loosdrecht AA, de Witte T, Cazzola M; European Leukemia Net. Diagnosis and treatment of primary myelodysplastic syndromes in adults: recommendations from the European LeukemiaNet. Blood. 2013 Oct 24;122(17):2943-64. doi: 10.1182/blood-2013-03-492884. Epub 2013 Aug 26. PMID 23980065
- [Background] Meldi K, Qin T, Buchi F, Droin N, Sotzen J, Micol JB, Selimoglu-Buet D, Masala E, Allione B, Gioia D, Poloni A, Lunghi M, Solary E, Abdel-Wahab O, Santini V, Figueroa ME. Specific molecular signatures predict decitabine response in chronic myelomonocytic leukemia. J Clin Invest. 2015 May;125(5):1857-72. doi: 10.1172/JCI78752. Epub 2015 Mar 30. PMID 25822018
- [Background] Montalban-Bravo G, Garcia-Manero G. Myelodysplastic syndromes: 2018 update on diagnosis, risk-stratification and management. Am J Hematol. 2018 Jan;93(1):129-147. doi: 10.1002/ajh.24930. PMID 29214694
- [Background] Prebet T, Gore SD, Esterni B, Gardin C, Itzykson R, Thepot S, Dreyfus F, Rauzy OB, Recher C, Ades L, Quesnel B, Beach CL, Fenaux P, Vey N. Outcome of high-risk myelodysplastic syndrome after azacitidine treatment failure. J Clin Oncol. 2011 Aug 20;29(24):3322-7. doi: 10.1200/JCO.2011.35.8135. Epub 2011 Jul 25. PMID 21788559
- [Background] Prebet T, Charbonnier A, Gelsi-Boyer V, Mozziconacci MJ, Blaise D, Vey N. Lenalidomide treatment for patients with myelodysplastic syndrome and low blast count acute myeloid leukemia after azacitidine failure. Leuk Lymphoma. 2013 Jul;54(7):1538-40. doi: 10.3109/10428194.2012.744455. Epub 2012 Nov 29. No abstract available. PMID 23110702
- [Background] Quesnel B, Guillerm G, Vereecque R, Wattel E, Preudhomme C, Bauters F, Vanrumbeke M, Fenaux P. Methylation of the p15(INK4b) gene in myelodysplastic syndromes is frequent and acquired during disease progression. Blood. 1998 Apr 15;91(8):2985-90. PMID 9531610
- [Background] Roboz GJ, Montesinos P, Selleslag D, Wei A, Jang JH, Falantes J, Voso MT, Sayar H, Porkka K, Marlton P, Almeida A, Mohan S, Ravandi F, Garcia-Manero G, Skikne B, Kantarjian H. Design of the randomized, Phase III, QUAZAR AML Maintenance trial of CC-486 (oral azacitidine) maintenance therapy in acute myeloid leukemia. Future Oncol. 2016 Feb;12(3):293-302. doi: 10.2217/fon.15.326. Epub 2016 Jan 19. PMID 26785287
- [Background] Santini V, Fenaux P, Mufti GJ, Hellstrom-Lindberg E, Silverman LR, List A, Gore SD, Seymour JF, Backstrom J, Beach CL. Management and supportive care measures for adverse events in patients with myelodysplastic syndromes treated with azacitidine*. Eur J Haematol. 2010 Aug;85(2):130-8. doi: 10.1111/j.1600-0609.2010.01456.x. Epub 2010 Apr 12. PMID 20394651
- [Background] Santini V, Prebet T, Fenaux P, Gattermann N, Nilsson L, Pfeilstocker M, Vyas P, List AF. Minimizing risk of hypomethylating agent failure in patients with higher-risk MDS and practical management recommendations. Leuk Res. 2014 Dec;38(12):1381-91. doi: 10.1016/j.leukres.2014.09.008. Epub 2014 Sep 22. PMID 25444075
- [Background] Santini V. How I treat MDS after hypomethylating agent failure. Blood. 2019 Feb 7;133(6):521-529. doi: 10.1182/blood-2018-03-785915. Epub 2018 Dec 13. PMID 30545832
- [Background] Shen L, Kantarjian H, Guo Y, Lin E, Shan J, Huang X, Berry D, Ahmed S, Zhu W, Pierce S, Kondo Y, Oki Y, Jelinek J, Saba H, Estey E, Issa JP. DNA methylation predicts survival and response to therapy in patients with myelodysplastic syndromes. J Clin Oncol. 2010 Feb 1;28(4):605-13. doi: 10.1200/JCO.2009.23.4781. Epub 2009 Dec 28. PMID 20038729
- [Background] Silverman LR, Demakos EP, Peterson BL, Kornblith AB, Holland JC, Odchimar-Reissig R, Stone RM, Nelson D, Powell BL, DeCastro CM, Ellerton J, Larson RA, Schiffer CA, Holland JF. Randomized controlled trial of azacitidine in patients with the myelodysplastic syndrome: a study of the cancer and leukemia group B. J Clin Oncol. 2002 May 15;20(10):2429-40. doi: 10.1200/JCO.2002.04.117. PMID 12011120
- [Background] Silverman LR, Fenaux P, Mufti GJ, Santini V, Hellstrom-Lindberg E, Gattermann N, Sanz G, List AF, Gore SD, Seymour JF. Continued azacitidine therapy beyond time of first response improves quality of response in patients with higher-risk myelodysplastic syndromes. Cancer. 2011 Jun 15;117(12):2697-702. doi: 10.1002/cncr.25774. Epub 2011 Jan 10. PMID 21656747
- [Background] Vardiman JW, Thiele J, Arber DA, Brunning RD, Borowitz MJ, Porwit A, Harris NL, Le Beau MM, Hellstrom-Lindberg E, Tefferi A, Bloomfield CD. The 2008 revision of the World Health Organization (WHO) classification of myeloid neoplasms and acute leukemia: rationale and important changes. Blood. 2009 Jul 30;114(5):937-51. doi: 10.1182/blood-2009-03-209262. Epub 2009 Apr 8. PMID 19357394
- [Background] Zeidan AM, Stahl M, Hu X, Wang R, Huntington SF, Podoltsev NA, Gore SD, Ma X, Davidoff AJ. Long-term survival of older patients with MDS treated with HMA therapy without subsequent stem cell transplantation. Blood. 2018 Feb 15;131(7):818-821. doi: 10.1182/blood-2017-10-811729. Epub 2017 Dec 19. No abstract available. PMID 29259002